CLINICAL TRIAL: NCT06375824
Title: Bufei Recipe Reduces the Incidence Rate of COPD: A Multicenter, Randomized, Double Blind, Placebo Controlled Study
Brief Title: Bufei Recipe Reduces the Incidence Rate of COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: West China Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for Pre-COPD
Record Dates: First submitted 2024-04-02; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Preserved Ratio Impaired Spirometry
Keywords: Bufei Recipe; PRISm; incidence rate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bufei Recipe (Experimental): Bu Fei Fang: Roasted Astragalus, Codonopsis pilosula, Walnut kernels, Sichuan Fritillaria, Angelica sinensis, Stir fried Purple Su Zi, Honey Baibu, Roasted Purple Aster, etc. Take 1 dose daily, 5 days a week.
  Interventions: Drug: Bufei Recipe
- Bufei Recipe placebo (Placebo Comparator): The placebo was prepared using 5% of the drug, with color, odor, taste, appearance, and weight similar to the experimental group drug, and packaging consistent with the experimental group drug.
  Interventions: Drug: Bufei Recipe placebo

INTERVENTIONS:
Drug: Bufei Recipe — Bufei Recipe: Roasted Astragalus, Codonopsis pilosula, Walnut kernels, Sichuan Fritillaria, Angelica sinensis, Stir fried Purple Su Zi, Honey Baibu, Roasted Purple Aster, etc. Take 1 dose daily, 5 days a week.
  Arms: Bufei Recipe
Drug: Bufei Recipe placebo — The placebo was prepared using 5% of the drug, with color, odor, taste, appearance, and weight similar to the experimental group drug, and packaging consistent with the experimental group drug.
  Arms: Bufei Recipe placebo

SUMMARY:
Establish early TCM prevention and treatment program to reduce the incidence rate of COPD.

DETAILED DESCRIPTION:
Taking PRISM patients with impaired lung function at the early stage of COPD retention ratio as the research object, and aiming at the key problems such as the lack of prevention and treatment plan, a two-year randomized double-blind placebo controlled clinical study of Bufei Fang was carried out to establish the early stage TCM prevention and treatment plan to reduce the incidence rate of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Risk factors for chronic obstructive pulmonary disease. Having one item from a, b, and c (risk factors will be further optimized based on the screening results of high-risk populations):

   1. smoking history (including previous and current smokers);
   2. 1 year or more of exposure to dust or chemical toxins;
   3. Indoor air pollution for 1 year or more (use of contaminated fuels, passive smoking, exposure) Oil fumes, etc.
2. Have a history of chronic bronchitis and/or emphysema, and have one of the following chronic respiratory symptoms:

   1. Cough (more than 3 months per year, continuous for 2 years or more);
   2. Coughing phlegm (more than 3 months per year, continuous for 2 years or more);
   3. Difficulty breathing (more than 3 months per year, continuous for 2 years or more).
3. The lung function test meets the following criteria: forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ≥ 70% and FEV1 accounting for%<80% of the expected value.
4. Meets the diagnostic criteria for lung qi deficiency syndrome.
5. Age range from 18 to 80 years old.
6. Voluntarily participate in the study and sign an informed consent form.

Exclusion Criteria:

* Pregnant and planned pregnancy, lactating women.
* Dementia and various mental illness patients.
* Other diseases with chronic cough, sputum production, or difficulty breathing.
* Merge tumors.
* Merge severe cardiovascular and cerebrovascular diseases.
* Concomitant severe liver and kidney diseases.
* Participants in clinical trials of other drugs.
* Allergies to intervention drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of COPD | Change from baseline in the number of people with COPD at month 24.
  Incidence rate of COPD

SECONDARY OUTCOMES:
FVC | Change from baseline in FVC at months 12 and 24.
  Forced Vital Capacity (FVC) was mainly used for lung function evaluation
FEV1 | Change from baseline in FEV1 at months 12 and 24.
  Forced Expiratory Volume in One Second (FEV1) was mainly used for lung function evaluation
FEV1% pred | Change from baseline in FEV1% pred at months 12 and 24.
  Percentage of Forced Expiratory Volume in One Second to Predicted Value (FEV1% pred) was mainly used for lung function evaluation
FEV1/FVC | Change from baseline in FEV1/FVC at months 12 and 24.
  Forced Expiratory Volume in One Second / Forced Vital Capacity (FEV1/FVC) was mainly used for lung function evaluation
IPAG-Q | Change from baseline in IPAG-Q score at months 6, 12, 18, and 24.
  International Primary Airway Health Organization Questionnaire (IPAG-Q) was mainly used for chronic obstructive pulmonary screening score evaluation.
LFQ | Change from baseline in LFQ score at months 6, 12, 18, and 24.
  Lung Function Questionnaire (LFQ) was mainly used for chronic obstructive pulmonary screening score evaluation.
COPD-PS | Change from baseline in COPD-PS score at months 6, 12, 18, and 24.
  Chronic Obstructive Pulmonary Disease Population Screening Questionnaire (COPD-PS) was mainly used for chronic obstructive pulmonary screening score evaluation.
CAT | Change from baseline in CAT score at months 6, 12, 18, and 24.
  Chronic Obstructive Pulmonary Disease Assessment (CAT) was mainly used for quality of life evaluation.
SF-36 | Change from baseline in SF-36 score at months 6, 12, 18, and 24.
  Health Survey Brief (SF-36) was mainly used for quality of life evaluation.
Clinical symptoms | Change from baseline in clinical symptom assessment questionnaire score at months 6, 12, 18, and 24.
  The assessment will be done through a clinical symptom assessment questionnaire. Clinical symptoms assessed in this study include cough, sputum, wheezing, chest tightness, shortness of breath, malaise and cyanosis. Each symptom or sign will receive a score of 0-3, with higher scores indicating greater severity of the condition.
Biochemical indicators | Change from baseline in biochemical indicators at month 12 and 24.
  Serum levels of TNF- α, IL-1, IL-6, immunoglobulin and renal connexin, prolyl peptidase, heme oxygenase-1, superoxide dismutase, glutathione peroxidase and angiotensin-converting enzyme were measured. All indicators were measured in ng/ml.

IPD SHARING:
Plan to Share IPD: No